CLINICAL TRIAL: NCT05369455
Title: Impact of Ultrasound Guided Erector Spine Plane & Caudal Block For Postoperative Analgesia In Pediatric Lower Limb Surgeries
Brief Title: Erector Spinae Plane Block in Pediatric Lower Limb Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Wafaa Madhy Atia Abdelwahed, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 35040/11/21
Record Dates: First submitted 2022-04-23; First posted 2022-05-11 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Efficacy of Erector Spinae Plane Block in Lower Limb Surgery in Pediatric
Keywords: erector spinae -block-pediatric -lower limb

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: neither investigator nor outcome assessors know which block patient had received
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): group of ultrasound guided Erector spine plane block:
  Interventions: Procedure: erector spinae plane block
- group 2 (Active Comparator): group of ultrasound guided Caudal block:
  Interventions: Procedure: ultrasound guided caudal block

INTERVENTIONS:
Procedure: erector spinae plane block — determine the efficacy and safety of ultra-sound guided erector spine plane block for providing postoperative analgesia in pediatric patients scheduled for lower limb surgeries as regard pain score , duration of analgesia and total postoperative analgesic requirement as a primary outcome as well as their safety as regard hemodynamics, adverse events local complications as secondary outcomes.
  Arms: group 1
Procedure: ultrasound guided caudal block — determine the efficacy and safety of ultra-sound guided caudal block for providing postoperative analgesia in pediatric patients scheduled for lower limb surgeries as regard pain score , duration of analgesia and total postoperative analgesic requirement as a primary outcome as well as their safety as regard hemodynamics, adverse events local complications as secondary outcomes.
  Arms: group 2

SUMMARY:
Anesthesia will be induced in all patients using Fentanyl 1µg,propofol 2mg/kg and cisatracurium 0.15 mg/kg IV to facilitate endotracheal intubation, maintenance of anaesthesia afterward will be achieved by isoflurane1.5-2% in oxygen and air mixture, cisatracurium0.03 mg/kg.

In both groups , ultrasound guided block will be performed by an experienced anesthesiologist who has no subsequent role in the study after induction of anesthesia and before starting of surgery in lateral position, sterilized and covered with sterile sheets. Aseptic precautions is taken by wearing sterile gowns and gloves A sterile preparation of the ultrasound probe is obligatory. Outcome parameters will be assessed by another anesthesiologist blinded to the groups of assignment.

Group 1: group of ultrasound guided Erector spine plane block:

Group 11: group of ultrasound guided Cauda block:

DETAILED DESCRIPTION:
Ethical considerations:

* After approval from institutional ethics committee, an informed consent will be obtained from all parents of participants in this research. All data of patients will be confidential with secret codes and private file for each patient, and all given data will be used for the current medical research only.
* Any unexpected risks appear during the course of the research will be cleared to the participants and ethical committee on time and proper measures will be taken to overcome or minimize these risks Patients will be randomized into two equal groups at a ratio of 1:1 to receive either Erector spine plane block (Group I n= 25) or Caudal block (Group II n= 25).

Randomization will be performed using sealed opaque envelopes indicating the group of assignment. A blinded nurse, who will not participate in the study or data collection, read the number contained in the envelope and made group assignments.

A preoperative evaluation in form of history taking, clinical examination and routine laboratory investigations, On arrival to the operating room, an intravenous (IV) cannula 24-22 gauge will be inserted and standard monitoring in terms of electrocardiogram (ECG), non-invasive blood pressure, capnograph and pulse oximeter for oxygen saturation (SpO2) will be connected to each participants. Patient received ,05mg midazolam and 4 mg ondansetron.

Anesthesia will be induced in all patients using Fentanyl 1µg,propofol 2mg/kg and cisatracurium 0.15 mg/kg IV to facilitate endotracheal intubation, maintenance of anaesthesia afterward will be achieved by isoflurane1.5-2% in oxygen and air mixture, cisatracurium0.03 mg/kg.

In both groups , ultrasound guided block will be performed by an experienced anesthesiologist who has no subsequent role in the study after induction of anesthesia and before starting of surgery in lateral position, sterilized and covered with sterile sheets. Aseptic precautions is taken by wearing sterile gowns and gloves A sterile preparation of the ultrasound probe is obligatory. Outcome parameters will be assessed by another anesthesiologist blinded to the groups of assignment.

Group 1: Technique of ultrasound guided Erector spine plane block:

The pa¬tient will be placed in in left lateral decubitus and the ultrasound-guided ESP block was performed at the(T12-L4) level on the left side.A 18_20 needle was inserted with the bevel in cephalo- caudal direction and 0.5 ml Kg of 0.25% Bupivacaine were injected Group 11: Technique of ultrasound guided Cauda block: With the patient in the left lateral decubitus position and the hips and knees flexed, the sacral hiatus can be identified using ultrasound First of all, the posterior superior iliac spines are palpated via anatomical landmarks, the line between both spines representing the base of an equilateral triangle the tip of which indicates the position of the sacral hiatus. The sacro coccygeal ligament can be palpated between the two sacral cornua, which is where the needle should penetrate the skin at an approximate 45 angle. Once the ligament has been passed, a flatter angle is adjusted by descending the needle before it can be advanced to the correct final position. Local anesthesia 0.5 ml Kg of 0.25% Bupivacaine were injected. Before application of local anesthetic , cautious aspiration or passive drainage is required to rule out an inadvertent intravascular or spinal needle location. Ultrasound guidance, by comparison ,offers two key advantages: it helps to identify small anatomical structures, and allows the spread of the local anesthetic to be seen by placing it longitudinally in a position slightly Para median to the lumbar spine .

ELIGIBILITY:
Inclusion Criteria:

* aged 2-15years old,
* classified by the American society of anesthesiologists as ASA I and II
* who will be scheduled for elective lower limb surgery will be enrolled in our study.

Exclusion Criteria:

* Parents refusal,

  * spine or chest wall deformity,
  * coagulation disorders, ,
  * known respiratory and cardiac disorders, renal or hepatic insufficiency
  * known allergy to study drugs, uncooperative patients.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
pain score | in first 24 hours postoperatively
  pain will be assessed using Face, Legs, Activity, Cry, and Consolability (FLACC) or Numeric Rating Scale (NRS) scores

SECONDARY OUTCOMES:
total postoperative analgesic requirement | first 24 hours postoperatively
  amount of postoperative analgesia (non steroidal )

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, Egypt